CLINICAL TRIAL: NCT01941550
Title: Neoadjuvant Chemotherapy With Cabazitaxel in High Risk Prostate Cancer Patients Prior to Radical Prostatectomy
Brief Title: Neoadjuvant Chemotherapy With Cabazitaxel
Acronym: CLUBNET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left the site. Site closed.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-005
Record Dates: First submitted 2013-07-22; First posted 2013-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: High-Risk Cancer
Keywords: untreated, high risk prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel chemotherapy (Other): Patients undergo 6 cycles Cabazitaxel chemotherapy. Cabazitaxel suspension is given once per cycle as infusion intravenously, 1 mg/square meter.
  For max. 6 times at all.
  Interventions: Drug: Cabazitaxel chemotherapy

INTERVENTIONS:
Drug: Cabazitaxel chemotherapy — given in 6 cycles
  Other Names: Jevtana L01CD04

SUMMARY:
This study is aimed at evaluating the efficacy regarding the response rate and metastasis-free survival time of cabazitaxel as a neoadjuvant treatment in patients with high risk prostate cancer.

DETAILED DESCRIPTION:
Patients will be treated by 6 cycles of Cabazitaxel 25 mg/m2 every three weeks and extended radical prostatectomy and extended pelvic lymphadenectomy 4 weeks after completion of chemotherapy. Multiparametric MRI will be performed at baseline, after 3 cycles and after 6 cycles. If there will be evidence of clinical progression after 3rd cycle, patients can be removed from the study and given local therapy, including radical prostatectomy or external beam radiotherapy, at the discretion of the patient's physicians. If patients have evidence of response, they continue on treatment for a total of 6 cycles. If multiparametric MRI demonstrates stable disease an individual risk-benefit analysis has to be performed with regard to continuing or to stopping the neoadjuvant treatment since the definition stable disease includes patients with ≤ 20% tumour shrinkage or tumour progression

ELIGIBILITY:
Inclusion Criteria:

* Surgically resectable high risk prostate cancer with a 5-year relapse probability ≥ 60% according to the Kattan pre-operative nomogram (cancer 2009, 115: 1005-1010)

  * no prior therapy for prostate cancer such as androgen deprivation therapy, radiation therapy, or chemotherapy
  * ECOG performance status 0-1
* No evidence of active infection

  * Hemoglobin >9.0 g/dL
  * Absolute neutrophil count >1.5 x 109/L,
  * Platelet count >100 x 109/L,
  * AST/SGOT and/or ALT/SGPT <2.5 x ULN;
  * Total bilirubin <1.0 x ULN,
  * Serum creatinine <1.5 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded)
  * Patient information and signature of informed consent
  * Male ≥ 18 years
  * Patients of reproductive age must take appropriate contraceptive precautions during and for 6 months after the end of their participation in the study

Exclusion Criteria:

* Evidence of lymph node, visceral or bone metastases

  * previous major intrapelvic surgery
  * previous radiation therapy to the small pelvis
  * any type of malignancies within the last 5 years except basalioma and non-muscle invasive urothelial cancer of the urinary bladder
  * previous chemotherapy with taxanes (docetaxel, paclitaxel, cabazitaxel) for any indication
  * Hypersensitivity to the active substance or to any of the excipients
  * Known or suspected brain metastases or leptomeningeal metastases
  * Active or symptomatic viral hepatitis or chronic liver disease
  * Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Complete pathological response rate | 5 years
  Primary endpoint: overall or cancer specific survival nor progression-free survival(PFS) in 5 years. Composite measurement.
  Key-parameters:
  * Complete pathohistological remission
  * Intra/perioperative compl.
  * PFS
  * Metastasis-FS
  * Biochemical, radiological, clinical PFS and androgen-deprivation FS
  * Objective progr. during cabazitaxel therapy (cab.th.) and post surgery
  * PSA response at the end of cab.th.
  * PSA progression after 12 w. of cab.th.
  * Percentage of pat. with undetectable PSA (<0.1 ng/ml) post surgery
  * Relationship between PSA kinetics, histol. response and MRI response
  * Role of pathohistol. parameters such as intraductal, cribriform growth patterns and effect on response
  * Immunohistochemical evaluation of prostate biopsy and radical prostatectomy specimens of markers potentially associated with chemoresistance: growth differentiation factor 15, surviving, beta-tubuline I & II, p53, bcl-2,
  * Measurement of the serum concentrations of free circulating mDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia, Germany